CLINICAL TRIAL: NCT03470181
Title: Applying Nutrient Drink Test in Understanding Pathophysiology of Cyclic Vomiting Syndrome
Brief Title: Applying Nutrient Drink Test in Understanding Pathophysiology of CVS
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Scott Gabbard, MD, Staff, The Cleveland Clinic
Other Study IDs: 17-1138
Record Dates: First submitted 2018-03-13; First posted 2018-03-19 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Cyclic Vomiting Syndrome
Keywords: Chronic nausea, intermittent vomiting, impaired accommodation
MeSH Terms: conditions — Familial cyclic vomiting syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with Diagnosed CVS: This cohort will consist of 15 current patients previously diagnosed with Cyclic Vomiting Syndrome.
  Interventions: Dietary Supplement: Ensure
- Healthy Volunteers: This cohort will consist of 15 healthy volunteers, with no history of Cyclic Vomiting.
  Interventions: Dietary Supplement: Ensure

INTERVENTIONS:
Dietary Supplement: Ensure — Participants will perform a Nutrient Drink Test. This consists of drinking 125mL of liquid Ensure four times, at five-minute intervals.

SUMMARY:
Cyclic vomiting syndrome is a disorder characterized by nausea and vomiting, separated by periods without any symptoms. There is very little research on this field at this point and most doctors do not fully understand the disorder. The goal of this study is to assess how the stomach empties food. Participants will be asked to participate in this study because either (a) they have been diagnosed and/or treated for cyclic vomiting syndrome in the past, or (b) they are physically healthy. The study seeks to compare how a healthy person's stomach empties to how the stomach of someone with cyclic vomiting disorder empties.

DETAILED DESCRIPTION:
Up to 14% of unexplained vomiting in adults is attributed to an under recognized and often misdiagnosed disorder termed cyclic vomiting syndrome (CVS). As CVS is better understood, gastroenterologists are increasingly recognizing the importance of timely diagnosis and early management for this chronic and debilitating disorder. Currently, the only gold standard diagnostic strategy involves evaluating clinical criteria set by the Rome Foundation, such as vomiting frequency and duration of episodes. Outside of these subjective criteria, no definitive and objective diagnostic strategy for cyclic vomiting syndrome exists.

Developing diagnostic strategies has been difficult given the exact etiology of CVS is still unknown. One physiologic theory includes rapid gastric emptying (GE)-or a dumping-like syndrome related to impaired gastric accommodation. A retrospective analysis observed rapid gastric emptying by standard 4-hour scintigraphic gastric emptying study in 80% of subjects, suggesting a relationship with CVS and rapid GE. In turn, rapid emptying has been hypothesized to relate with abnormal gastric accommodation - the reflex allowing storage of food through increased fundic volume. This physiologic abnormality can be readily and easily measured using non-invasive tools, but have never been tested in CVS. To explore this further, we aim to determine if CVS patients have abnormal gastric accommodation measured by nutrient drink test.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Cyclic Vomiting (or Healthy Volunteer)
* Age 18 or greater

Exclusion Criteria:

* Age Under 18
* History of gastric surgery
* History of marijuana use
* History of Gastroparesis
* History of Diabetes mellitus II
* Upper endoscopy with known obstructive gastric disease
* Current pregnancy or lactation
* Active inflammatory bowel disease (Crohn's disease, Ulcerative colitis)
* Severe renal disease (GFR <15/dialysis dependent)
* Active malignancy (diagnosed in last 5 years)
* Allergy/intolerance to liquid Ensure®

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study seeks to enroll adult patients diagnosed with Cyclic Vomiting Syndrome, as well as healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated volume | Within 30 minutes of beginning the test.
  The amount of nutrient drink consumed before the participant reports feelings of unbearable fullness.

SECONDARY OUTCOMES:
Total Aggregate Symptom Score | Within 30 minutes of the beginning of the test
  Participant-Reported impressions of fullness, bloating, or abdominal pain, measures on 100mm visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Scott Gabbard, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No